CLINICAL TRIAL: NCT04147611
Title: Remote Microphone (RM) Technology in Children Using Bone Conduction Devices: A Comparative Study
Brief Title: Remote Microphone (RM) - A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Cochlear (Industry)
Responsible Party: Principal Investigator, Hillary A Snapp, Associate Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20190308
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Hearing Loss, Conductive
MeSH Terms: conditions — Hearing Loss, Conductive | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Remote Microphone (RM) Technology Group (Experimental): The RM technology group will limited to the pediatrics participants.
  Participants will be tested separately on the three following conditions:
  1. Bone Conduction Device (BAHA) only
  2. BAHA + Wireless Audio-Streaming Accessory
  3. BAHA + Digital Adaptive RM System
  Interventions: Device: BAHA; Device: Wireless Audio Streaming Accessory; Device: Digital Adaptive RM System
- Normal Hearing Controls (Active Comparator): The normal hearing controls will be limited to 15 adults.
  Participants will be tested separately on the six following conditions:
  1. Unaided
  2. Unilateral hearing aid with contralateral plug.
  3. Unilateral hearing aid + Digital Adaptive RM System (using Roger™, Sonova)
  4. Bone Conduction Device (BAHA) only
  5. BAHA + Wireless Audio-Streaming Accessory
  6. BAHA + Digital Adaptive RM System
  Interventions: Device: BAHA; Device: Wireless Audio Streaming Accessory; Device: Digital Adaptive RM System; Device: Hearing Aid

INTERVENTIONS:
Device: BAHA — Participant's pediatric bone conduction hearing device.
Device: Wireless Audio Streaming Accessory — Cochlear Corporation's Mini Microphone 2+ Wireless Audio Streaming Accessory is an accessory used to transmit speech and sound. It consists of a microphone and a transmitter that transfers the signal to a receiver that's connected to a hearing device.
Device: Digital Adaptive RM System — Sonova's Roger Digital Adaptive RM system is an accessory which can be connected to a compatible hearing aid. It offers an external microphone which streams signals directly to the connected hearing aid.
Device: Hearing Aid — Participant's unilateral hearing aid with contralateral plug.
  Arms: Normal Hearing Controls

SUMMARY:
The purpose of this investigation is to evaluate objective outcomes in pediatric bone conduction hearing device (often termed "BAHA") users with and without remote microphone (RM) technology. In this study, two remote microphone technologies will be evaluated to determine benefit in speech understanding in noise.

ELIGIBILITY:
Pediatric RM Technology Group:

Inclusion Criteria:

* English speaking pediatric conduction device users and their guardian/s will be included for study.
* We will include pediatric patients 5 years of age to 17 years of age who have a conductive or mixed unilateral or bilateral hearing loss with a minimum of a 30 decibels (dB) air-bone gap.

Exclusion Criteria:

- Participants who do not meet the described inclusion criteria.

Normal Hearing Controls:

Inclusion Criteria:

* Adults greater than18 years of age.
* Hearing thresholds < 25 dB 500 - 4,000 Hz.

Exclusion Criteria:

- Non-English speakers.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Snapp, AuD, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Kristine Harris, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Remote Microphone (RM) Technology Group: The RM technology group will limited to the pediatrics participants.
  Participants will be tested separately on the three following conditions:
  1. Bone Conduction Device (BAHA) only
  2. BAHA + Wireless Audio-Streaming Accessory
  3. BAHA + Digital Adaptive RM System
  BAHA: Participant's pediatric bone conduction hearing device.
  Wireless Audio Streaming Accessory: Cochlear Corporation's Mini Microphone 2+ Wireless Audio Streaming Accessory is an accessory used to transmit speech and sound. It consists of a microphone and a transmitter that transfers the signal to a receiver that's connected to a hearing device.
  Digital Adaptive RM System: Sonova's Roger Digital Adaptive RM system is an accessory which can be connected to a compatible hearing aid. It offers an external microphone which streams signals directly to the connected hearing aid.
- Normal Hearing Controls: The normal hearing controls will be limited to 15 adults.
  Participants will be tested separately on the six following conditions:
  1. Unaided
  2. Unilateral hearing aid with contralateral plug.
  3. Unilateral hearing aid + Digital Adaptive RM System (using Roger™, Sonova)
  4. Bone Conduction Device (BAHA) only
  5. BAHA + Wireless Audio-Streaming Accessory
  6. BAHA + Digital Adaptive RM System
  BAHA: Participant's pediatric bone conduction hearing device.
  Wireless Audio Streaming Accessory: Cochlear Corporation's Mini Microphone 2+ Wireless Audio Streaming Accessory is an accessory used to transmit speech and sound. It consists of a microphone and a transmitter that transfers the signal to a receiver that's connected to a hearing device.
  Digital Adaptive RM System: Sonova's Roger Digital Adaptive RM system is an accessory which can be connected to a compatible hearing aid. It offers an external microphone which streams signals directly to the connected hearing aid.
  Hearing Aid: Participant's unilateral hearing aid with contralateral plug.
Period: Overall Study
Arm/Group | Remote Microphone (RM) Technology Group | Normal Hearing Controls
Started | 9 | 13
Completed | 9 | 12
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote Microphone (RM) Technology Group | Normal Hearing Controls | Total
Number analyzed (Participants) | 9 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.67 (3.54) | 27.83 (4.73) | 20.90 (9.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Correct Word Responses
Description: Percentage of correct word responses as assessed via the Pediatric AZBio Sentence List test at -10 decibels (dB) signal to noise ratio. The total score ranges from 0-100% with the higher score indicating increased listening in noise performance.
Time Frame: 2 hours
Population: Data is provided for all participants who completed the study.
Measure: Mean (Standard Deviation); unit: percentage of correct word responses
Arm/Group | Remote Microphone (RM) Technology Group | Normal Hearing Controls
Number analyzed (Participants) | 9 | 12
percentage of correct word responses
  Bone Conduction Device (BCD) / Baha BCD only | 2.21 (3.6) | 0.1 (0.4)
  BCD/Baha BCD and Remote Microphone (RM) | 71.7 (24.3) | 87.9 (8.7)
  BCD/Baha BCD, RM, and Digital RM | 1.5 (2.2) | 11.2 (13.9)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Remote Microphone (RM) Technology Group | Normal Hearing Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT04147611/Prot_SAP_000.pdf